CLINICAL TRIAL: NCT01431209
Title: A Phase 2 Multicenter, Investigator Initiated Study of Oral Ruxolitinib Phosphate for the Treatment of Relapsed or Refractory Diffuse Large B-Cell and Peripheral T-Cell Non-Hodgkin Lymphoma
Brief Title: Ruxolitinib Phosphate to Treat Diffuse Large B-Cell or Peripheral T-Cell Non-Hodgkin Lymphoma After Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0283-11-FB; NCI-2011-02733 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2011-09-05; First posted 2011-09-09 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Mature T- and NK-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ruxolitinib phosphate) (Experimental): Patients receive ruxolitinib phosphate PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Ruxolitinib Phosphate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi

SUMMARY:
This phase II trial studies how well ruxolitinib phosphate works in treating patients with diffuse large B-cell or peripheral T-cell non-Hodgkin lymphoma that has returned (relapsed) or that does not respond to treatment (refractory) after donor stem cell transplant. Ruxolitinib phosphate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the overall response rate (ORR) of subjects with relapsed diffuse large B-cell lymphoma (DLBCL) and peripheral T-cell lymphoma (PTCL) who are relapsed or refractory to front-line treatment and ineligible for stem cell transplantation or have recurrent disease after stem cell transplantation to oral ruxolitinib (ruxolitinib phosphate).

SECONDARY OBJECTIVES:

I. Evaluate safety of oral ruxolitinib in subjects with DLBCL and PTCL. II. Determine progression-free survival (PFS), duration of response, and overall response (OS) in subjects with DLBCL and PTCL.

TERTIARY OBJECTIVES:

I. Explore the relationship between responses to oral ruxolitinib and alterations in gene expression profiling (GEP) signatures as well as biomarker immunophenotypic changes related to JAK2/STAT3, NF-kB, PI3K/AKT, and mTOR pathways.

II. Evaluate potential effect of oral ruxolitinib exposure on JAK2/STAT3 pathway inhibition in serial tumor samples.

OUTLINE:

Patients receive ruxolitinib phosphate orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically documented relapsed or refractory disease, with a diagnosis of one of the following lymphoid malignancies: diffuse large B-cell lymphoma, peripheral T-cell lymphoma (any subtype); subjects must have received at least one prior systemic chemotherapy and must have either received an autologous stem cell transplant, refused or been deemed ineligible for an autologous stem cell transplant
* Subjects must be willing and able to have a fresh tumor biopsy prior to start of study treatment for research evaluations and cohort categorizing; Note: if insufficient fresh tissue is obtained to provide sub-classification for cohorts, then tissue material from a previous relapse biopsy and/or original diagnostic block may be requested to meet this criterion
* Subjects must have measurable lesions (at least one target lesion measuring 2 cm in diameter) by computerized tomography (CT) scan, and/or measurable lymphoma cutaneous lesions of any size
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count >= 75,000/mm^3
* Hemoglobin >= 8.0 g/dL
* Serum creatinine =< 2.0 g/dL or calculated creatinine clearance >= 60 mL/min (Cockcroft-Gault method)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal (ULN) or =< 5 x ULN if liver involved by lymphoma
* Bilirubin < 2.0 x ULN unless subject has Gilbert's disease, low-grade hemolysis, or liver involvement with lymphoma
* At least 2 weeks since prior chemotherapy, biological therapy, radiation therapy, major surgery, other investigational, or anti-cancer therapy that is considered disease-directed and recovered from prior toxicities to grade 0-1 at least 2 weeks prior to investigational therapy
* Females will be either postmenopausal for at least 1 year or surgically sterile for at least 3 months; OR females of child-bearing potential must have a negative pregnancy test at screening and agree to take appropriate precautions to avoid pregnancy from screening until 3 months after their last dose of study medication
* Males must agree to take appropriate precautions to avoid fathering a child from screening until 3 months after their last dose of study medication
* Able to comprehend and willing to sign an informed consent form (ICF)

Exclusion Criteria:

* History of or active central nervous system (CNS) malignancy
* Allogeneic stem cell transplant within the last 6 months, or active-graft-versus-host disease following allogeneic transplant, or subjects currently on immunosuppressive therapy following allogeneic transplant
* Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements as judged by treating physician; subjects receiving antibiotics that are under control may be included in the study
* Pregnant or breastfeeding women
* Clinically symptomatic and uncontrolled cardiovascular disease
* History of myocardial infarction, severe/unstable angina, or symptomatic congestive heart failure, within the 6 months prior to study drug administration
* Current or recent history (< 21 days prior to start of treatment) of a clinically significant bacterial, viral, fungal, parasitic or mycobacterial infection
* History of other malignancy, with the exception of squamous cell carcinoma of the skin, basal cell carcinoma of the skin, cervical intraepithelial neoplasia, or other malignancies that have been in remission for at least 3 years
* Presence of a malabsorption syndrome possibly affecting drug absorption (e.g., Crohn's disease or chronic pancreatitis)
* Any prior or concomitant use of another JAK inhibitor
* Known active hepatitis B or C, or human immunodeficiency virus (HIV) infection
* Subjects who, in the opinion of the investigator, are unable or unlikely to comply with the dosing schedule and study evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-08-12 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, MBA, Principal Investigator — University of Nebraska
Locations (3):
- United States (3):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska

REFERENCES:
- [Derived] Wang C, Althof PA, Bi C, Zhang W, Bouska AC, Tian T, Zhang X, Jiang N, Yu G, Cheng H, Iqbal J, Vose JM, Sanmann JN, Fu K. A novel MYC-non-IG fusion in refractory diffuse large B-cell lymphoma. Br J Haematol. 2021 Jun;193(5):1001-1004. doi: 10.1111/bjh.17255. Epub 2021 May 3. No abstract available. PMID 33942298

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Evaluable population - Subjects who had completed 2 cycles of therapy with response assessments or progressed before the evaluation of the primary endpoint.
  Primary endpoint The primary objective of the study is to evaluate subject overall response rate (ORR) after 6 cycles for each of the subject cohorts. The description provided in this section includes the primary analyses for the primary objective.
Pre-assignment Details: For this study 71 subjects were screened and consented for the study. Nine were considered ineligible by the principal investigator and were not treated and removed from the study. Two other subjects were also not included in the data analysis. One withdrew consent prior to treatment. One was determined to have disease progression before treatment started.
Groups:
- Diffuse Large B-cell Lymphoma (DLBCL); Peripheral T-cell Non-Hodgkin Lymphoma (PTCL): Patients receive ruxolitinib phosphate PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  Ruxolitinib Phosphate: Given PO
Period: Overall Study
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Non-Hodgkin Lymphoma (PTCL)
Started | 47 | 13
Completed | 43 | 12
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Non-Hodgkin Lymphoma (PTCL) | Total
Number analyzed (Participants) | 47 | 13 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11) | 66 (13) | 65 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 5 | 23
  Male | 29 | 8 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  White | 40 | 12 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 47 | 13 | 60

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Number of patients achieving overall response rate
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Non-Hodgkin Lymphoma (PTCL)
Number analyzed (Participants) | 47 | 13
Participants
  Complete Response | 1 | 1
  Partial Response | 3 | 1
  Stable disease | 5 | 3
  Progressive disease | 34 | 7
  Not assessed | 4 | 1

2. Secondary Outcome: Overall Survival (OS)
Description: The Kaplan-Meier method will be used to estimate the median OS time and its 95% CI.
Time Frame: From the date of start of treatment to date of death due to any cause, assessed up to 60 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Non-Hodgkin Lymphoma (PTCL)
Number analyzed (Participants) | 47 | 13
Months | 5.9 [3.3 to 14.3] | 6.9 [3.8 to 24.3]

3. Secondary Outcome: Progression-free Survival
Description: The Kaplan-Meier method will be used to estimate the median PFS time and its 95% CI.
Time Frame: From the date of start of treatment to the date of event defined as the first documented progression or death due to any cause, assessed up to 60 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Non-Hodgkin Lymphoma (PTCL)
Number analyzed (Participants) | 47 | 13
Months | 1.8 [1.1 to 1.8] | 2.2 [0.9 to 4.6]

ADVERSE EVENTS:
Time Frame: Adverse Event monitoring should be continued for at least 30 days following the last dose of study treatment. Since this treatment trial was for relapsed or refractory disease in subjects, subjects were allowed to continue study treatment as long as they received benefit and met not reason for study discontinuation. The last subject remained on treatment for 7 1/2 years.
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Non-Hodgkin Lymphoma (PTCL)
All-Cause Mortality (participants affected / at risk) | 31/47 | 11/13
Serious Adverse Events (participants affected / at risk) | 22/47 | 7/13
Other Adverse Events (participants affected / at risk) | 43/47 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-cell Lymphoma (DLBCL) (N=47) | Peripheral T-cell Non-Hodgkin Lymphoma (PTCL) (N=13)
Fever (General disorders) | 6 | 3
Infections and infestiations - Other (Infections and infestations) | 1 | 0 — Thrush
Respiratory disorder- other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — pneumonia
Anemia (Blood and lymphatic system disorders) | 1 | 2
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
fatigue (General disorders) | 0 | 1
febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
hypernatremia (Metabolism and nutrition disorders) | 0 | 1
hyponatremia (Metabolism and nutrition disorders) | 0 | 1
hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
hypotension (Vascular disorders) | 1 | 1
Injury, procedural - Other (Injury, poisoning and procedural complications) | 0 | 1 — right shin wound
lung infection (Infections and infestations) | 2 | 1
Musculoskeletal, Other (Musculoskeletal and connective tissue disorders) | 1 | 1 — body weakness
pleuritc pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
sepsis (Infections and infestations) | 4 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
thromboembolic event (Vascular disorders) | 3 | 0
Acute kidney injury (Injury, poisoning and procedural complications) | 2 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
ileus (Gastrointestinal disorders) | 2 | 0
Infections - Other (Infections and infestations) | 1 | 0 — pneumocystis pneumonia
infections - Other (Infections and infestations) | 0 | 1 — respiratory syncytial virus
Infections - Other (Infections and infestations) | 0 | 1 — bacteremia
Other infection (Infections and infestations) | 0 | 1 — wound infection
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
sinus tachycardia (Cardiac disorders) | 2 | 0
abdominal pain (Gastrointestinal disorders) | 1 | 0
anorexia (Metabolism and nutrition disorders) | 1 | 0
cardiac disorder, Other (Cardiac disorders) | 1 | 0 — cardiomyopathy
cognitive disturbance (Nervous system disorders) | 1 | 0
confusion (Psychiatric disorders) | 1 | 0
creatinine increased (Investigations) | 1 | 0
delirium (Psychiatric disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 1 | 0
dizziness (Nervous system disorders) | 1 | 0
fracture (Injury, poisoning and procedural complications) | 1 | 0
gait disturbance (General disorders) | 1 | 0
gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hepatobiliary - Other (Hepatobiliary disorders) | 1 | 0 — steatohepatitis
hypertension (Vascular disorders) | 1 | 0
Investigations (Investigations) | 1 | 0 — acute kidney injury
leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
lymphedema (Vascular disorders) | 1 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
platelet count decreased (Blood and lymphatic system disorders) | 1 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
seizure (Nervous system disorders) | 1 | 0
skin infection (Skin and subcutaneous tissue disorders) | 1 | 0
syncope (Nervous system disorders) | 1 | 0
tumor lysis syndome (Metabolism and nutrition disorders) | 1 | 0
upper respiratory infection (Infections and infestations) | 1 | 0
vomiting (Gastrointestinal disorders) | 1 | 0
wound infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-cell Lymphoma (DLBCL) (N=47) | Peripheral T-cell Non-Hodgkin Lymphoma (PTCL) (N=13)
Respiratory, thoracic and mediastinal disorder - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — actelectasis
fatigue (General disorders) | 2 | 2
hyponatremia (Metabolism and nutrition disorders) | 0 | 2
anemia (Blood and lymphatic system disorders) | 11 | 1
apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
fever (General disorders) | 2 | 1
hypercalcemia (Metabolism and nutrition disorders) | 2 | 1
hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1
hypotension (Vascular disorders) | 2 | 1
lung infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1
lymphocyte count decreased (Investigations) | 4 | 1
malaise (General disorders) | 0 | 1
Musculoskeletal, Other (Musculoskeletal and connective tissue disorders) | 0 | 1 — facial and neck swelling
nausea (Gastrointestinal disorders) | 1 | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
platelet count decreased (Investigations) | 5 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
neutrophil count decreased (Investigations) | 4 | 0
sepsis (Infections and infestations) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT01431209/Prot_SAP_000.pdf